CLINICAL TRIAL: NCT04221971
Title: Clinical Study of Natural Killer Cell Infusion in Patients With Acute Myeloid Leukemia
Brief Title: NK Cell Infusion for Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: The University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, President, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019PHD005-01
Record Dates: First submitted 2019-12-02; First posted 2020-01-09 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AML patients with NK cells infusion (Experimental): The relapsed/refractory AML patient received Flu+CTX (Flu 25mg/m2 (-6d to -2d)，CTX 1.0g/m2 (-6d to -5d) and haploidentical NK cells infusion postchemotherapy for at least 48 hours. NK cell dose was over 1+E07/ kg with 3 consecutive infusions. NK cells infusion interval was 1 day.
  Interventions: Drug: chemotherapy combined with NK cells infusion

INTERVENTIONS:
Drug: chemotherapy combined with NK cells infusion — chemotherapy combined with NK cells infusion
  Other Names: cyclophosphamide (Cy, 1000 mg/m2/day, day -6 to -5), and fludarabine (Flu, 25 mg/m2/day, day -6 to -2)

SUMMARY:
Natural killer (NK) cells exert antitumor effects via their cytotoxic and cytokine-secreting capacity without present of clinical symptoms. In recent years, with the continuous advancement of in vitro expansion methods, the application of good quality management technology, NK cells could be clinical grade expanded without the need for pre-purification, feeder-free, and serum-free culture. In this clinical trial the investigators want to demonstrate the safety and efficacy chemotherapy combined with donor-derived in vitro activated NK cells infusion for high risk AML patients.

DETAILED DESCRIPTION:
Despite improvements in new drugs and allogeneic stem cell transplantation (allo-SCT), relapse remains a problem for patients with acute myeloid leukemia (AML). Natural killer (NK) cells exert antitumor effects via their cytotoxic and cytokine-secreting capacity without present of clinical symptoms.

In recent years, with the continuous advancement of in vitro expansion methods, the application of good quality management technology (GMP technology), NK cells could be clinical grade expanded without the need for pre-purification, feeder-free, and serum-free culture. Preclinical studies have confirmed that adoptive infusion expanded and activated NK cells can specifically recognize and kill tumor cells in mice without causing GVHD, which is a safe and effective treatment.

Therefore, in this clinical trial the investigators want to enroll patients with acute AML (excluding APL) who are continued to be unresolved, or relapsed after remission, or continued to be MRD-positive after induction and consolidation according to NCCN standard chemotherapy regimen. Chemotherapy was combined with donor-derived in vitro activated NK cells infusion to evaluate the safety and effectiveness effect of NK cells and to explore the dynamics of NK in vivo after adoptive infusion.

ELIGIBILITY:
Inclusion Criteria:

1. AML patients receiving standard NCCN induction and consolidation chemotherapy;
2. Age> = 18 years old;
3. Relapsed and refractory AML: continued non-remission after induction and consolidation chemotherapy with NCCN standard protocol, or relapse after remission, or continued MRD positive;
4. MDS-RAEB, MDS-AML, MPD-AML;
5. ECOG≤3;
6. No serious organ dysfunction within 2 weeks before treatment:

   1. Heart: no arrhythmia and LVEF≥50% and no pericardial effusion;
   2. Liver: liver function <2 times the upper limit of ALT and <1.5 times the upper limit of total bilirubin, no active hepatitis;
   3. Kidney: serum creatinine <1.5 mg / dl; or if serum creatinine exceeds the upper limit, serum creatinine clearance should be CrCl> 50 ml / min;
   4. indoor fingertip blood oxygen saturation ≧ 92%;
7. Expected survival time ≥ 3 months;
8. The interval between re-induction therapy and NK cell therapy is at least 2 weeks, and the toxic and side effects of all induction remission treatments have disappeared; if the patient is receiving non-invasive chemotherapy, such as hydroxyurea, low-dose cytarabine, before receiving this program Should be discontinued before;
9. All patients and donors are willing to join this clinical trial and sign informed consent.

Exclusion Criteria:

1. Combined with a history of other malignant tumors <5 years (except cured skin basal cell carcinoma, cured cervical carcinoma in situ and gastrointestinal tumors confirmed to be cured by endoscopic mucosal resection);
2. Have received bone marrow or organ transplant;
3. Those who are allergic to the biological agents used in this treatment;
4. active infection;
5. Those who received other cell treatments such as DLI, CMV-CTL, EBV-CTL;
6. HBV carriers;
7. Patients with extramedullary recurrence;
8. Chest radiographic examination to determine patients with pulmonary inflammation;
9. Researchers do not consider it appropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Two months after NK treatment
  Closely monitor the patient's temperature, rash, BP, and other adverse reactions during the 48 hours after the infusion, and pay attention to acute and chronic GVHD; follow up once every 1-2 weeks within 6 months after the infusion, and review the blood count and biochemistry. Increase or decrease the relevant inspections and inspection frequencies as appropriate according to the condition;

SECONDARY OUTCOMES:
Number of participants acheived CR post NK treatment | One month after NK treatment
  To evaluate the CR rate 1 month after NK treatment
Monitor the metabolism, migration and reconstruction of NK cells in vivo post NK treatment | One month after NK treatment
  The number of NK cells were evaluated before and after the completion of the infusion.
Assess the cell count recovery time of peripheral blood in chemotherapy combined with NK infusion | Two months after NK treatment
  The blood count were evaluated closely before and after the completion of the infusion.
Number of participants relapsed post NK treatment | Every months after NK treatment within 1 year
  To evaluate the bone marrow status every months after NK treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, M.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No